CLINICAL TRIAL: NCT01319539
Title: Pre-surgical Evaluation of MK-2206 in Patients With Operable Invasive Breast Cancer
Brief Title: MK2206 in Treating Patients With Stage I, Stage II, or Stage III Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: terminated early, due to toxicity
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02513; NCI-2011-02513 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000696821 (Other: NCI); AECM-AAAF3912 (Other: Montefiore Medical Center - Moses Campus); 8740 (Other: CTEP); N01CM62204 (NIH); P30CA013330 (NIH)
Record Dates: First submitted 2011-03-18; First posted 2011-03-21 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Estrogen Receptor Negative; Estrogen Receptor Positive; HER2/Neu Negative; HER2/Neu Positive; Progesterone Receptor Negative; Progesterone Receptor Positive; Stage IA Breast Cancer; Stage IB Breast Cancer; Stage IIA Breast Cancer; Stage IIB Breast Cancer; Stage IIIA Breast Cancer; Stage IIIB Breast Cancer; Stage IIIC Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — MK 2206

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO on days -9 and -2, and undergo segmental resection or total mastectomy (therapeutic conventional surgery) on day 0. Patient samples will be processed for pharmacological study and laboratory biomarker analysis.
  Interventions: Drug: Akt Inhibitor MK2206; Procedure: Therapeutic Conventional Surgery; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Procedure: Therapeutic Conventional Surgery — Undergo surgery
Other: Pharmacological Study — Correlative studies
  Other Names: pharmacological studies
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studies how well Akt inhibitor MK2206 works in treating patients with stage I-III breast cancer that can be removed by surgery. Akt inhibitor MK2206 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess for a decrease in phosphorylated (phospho)-protein kinase B (Akt) (Ser^473) levels in tissue after a pre-surgical trial of weekly MK2206 (Akt inhibitor MK2206) (2 doses) in patients with operable invasive breast cancer.

SECONDARY OBJECTIVES:

I. To evaluate the effects of MK2206 on the immunohistochemical expression of other phosphatidylinositide 3-kinase (PI3K)/AKT pathway biomarkers on pre-and post-MK2206 tumor tissue, such as phospho-S6 kinase.

II. To assess modulation of PI3K/AKT signaling following MK2206 use with reverse-phase protein microarray analysis.

III. To explore whether phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutations demonstrate different modulation of PI3K/Akt-pathway signaling as compared to tumors with loss of phosphatase and tensin homolog (PTEN).

IV. To explore whether MK2206 alters PI3K/Akt pathway signaling differently in hormone receptor-positive/human epidermal growth factor receptor (HER)2-negative tumors, as compared to triple-negative or HER2-positive breast cancers.

V. To evaluate whether tumor proliferation, as measured by Ki-67 staining of breast tumor cells, is reduced in patients taking MK2206 pre-surgically and correlate Ki-67 modulation with changes in PI3K/AKT signaling.

VI. To determine safety and tolerability of MK2206 in patients with early-stage breast cancer.

VII. To collect fasting blood for evaluation of predictive markers of drug effect, such as markers in the insulin growth-factor receptor pathway (i.e., fasting insulin, c-peptide, insulin-like growth factor [IGF]-1, and IGF binding protein [BP]-1 and 3), as well as modulation of phospho-markers in peripheral blood mononuclear cells.

OUTLINE:

Patients receive Akt inhibitor MK2206 orally (PO) on days -9 and -2, and undergo segmental resection or total mastectomy on day 0.

After completion of study treatment, patients are followed up for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically-confirmed operable invasive breast cancer and have undergone core needle biopsy with an anticipated surgical resection for residual disease after enrollment
* Patients must have clinical stage I-III invasive breast (invasive tumor must be clinically at least >= T1c by radiograph or palpation)
* Patients must have available tissue from core biopsies for biomarker assessment; it is recommended that at least 4 cores be performed with 12 gauge (or smaller gauge) needles; this includes cores underneath ultrasound-guidance
* Patients are planning to undergo surgical treatment with either segmental resection or total mastectomy (required: 2 doses of weekly MK-2206 prior to surgery; the first dose will be at day -9 [+/- 1 day] and second dose at day -2 [+/- 1 day] in relation to surgery [day 0])
* Patients may have a history of contralateral breast cancer, provided there is no evidence of recurrence of the initial primary breast cancer
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Karnofsky >= 80%)
* Leukocytes >= 3,000/ul within 28 days of registration
* Platelets >= 100,000 /uL within 28 days of registration
* Hemoglobin (Hgb) >= 9 g/dL within 28 days of registration
* Creatinine =< 1.5 x upper limit of normal (ULN) within 28 days of registration
* Prothrombin time (PT), partial thromboplastin time (PTT) =< 1.2 x ULN within 28 days of registration
* Total bilirubin =< 1.5 x ULN within 28 days of registration
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x ULN within 28 days of registration
* Patients of childbearing potential must have a negative serum or urine pregnancy test beta-human chorionic gonadotropin (β-hCG) within 72 hours prior to receiving the first dose of study medication
* Women of childbearing potential and men must use two forms of contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, the patient should inform the treating physician immediately
* Patient must be able to swallow oral tablets
* Ability to understand and the willingness to sign a written informed consent document
* Patients must agree to biomarker assessment of pre-treatment diagnostic core biopsy tissue and the surgical resection tissue (i.e. excision or mastectomy); also, must agree to pre- and post-treatment fasting blood biomarker collection

Exclusion Criteria:

* Patients may not have any known evidence of distant metastatic disease (i.e., lung, liver, bone, or brain metastases) or locally recurrent breast cancer
* Patients with inflammatory breast cancer are not eligible
* Patients with prior chemotherapy or radiation therapy within 6 months of study entry are not eligible (i.e. patient who have received neoadjuvant therapy are not eligible)
* Patients may not be receiving any other investigational agents, including other inhibitors of PI3K, Akt, or mammalian target of rapamycin (mTOR)
* Men diagnosed with breast cancer
* Patients may not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-2206 used in the study
* Patients with known diabetes which is poorly controlled diabetes (hemoglobin A1c [HBA1C] >= 8%) should be excluded; if patient is taking metformin, must have been taking this medication for > 3 months, as metformin is thought to impact PI3K/Akt signaling
* Baseline corrected QT interval (QTc) > 470 msec will exclude patients from entry on study; patients with a baseline bundle branch block will be excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with MK2206
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kalinsky, Principal Investigator — Montefiore Medical Center - Moses Campus
Locations (3):
- United States (3):
  - Columbia University Medical Center, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 participants were enrolled between September 2011 and March 2013.
Groups:
- Treatment (Akt Inhibitor MK2206): Patients receive Akt inhibitor MK2206 PO on days -9 and -2, and undergo segmental resection or total mastectomy on day 0.
  Akt Inhibitor MK2206: Given PO
  Therapeutic Conventional Surgery: Undergo surgery
  Pharmacological Study: Correlative studies
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 7
  Non-Hispanic White | 4
  Non-Hispanic Black | 1
  Asian | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in pAKT Levels
Description: This is designed to evaluate response to therapy - comparing changes within group (example: invasive pre-MK-2206-treated core versus post-MK-2206-treated surgical tissue).
Time Frame: Baseline, 2 weeks (Day 0 - surgery)
Population: Of the 12 participants enrolled and received study treatment, there were 7 participants with evaluable matched core and surgical specimen tissue.
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 7
percentage of cells
  Core | 25 (29)
  Surgery | 0 (0)

2. Secondary Outcome: Change in pS6 Levels
Description: as for outcome 1
Time Frame: Baseline, 2 weeks (Day 0 - surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 7
percentage of cells
  Core | 41 (36)
  Surgery | 31 (32)

3. Secondary Outcome: Change in Ki-67 Expression
Description: as for outcome 1
Time Frame: Baseline, 2 weeks (Day 0 - surgery)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of cells
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 7
percentage of cells
  Core | 13 (23)
  Surgery | 12 (23)

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The definition of adverse event and/or serious adverse event, used to collect adverse event information, does not differ from the ClinicalTrials.gov definitions.
Groups:
- Treatment (MK2206) Dose Level 200mg; Treatment (MK2206) Dose Level 135mg; Treatment (MK2206) Dose Level 90mg: Patients receive Akt inhibitor MK2206 PO on days -9 and -2, and undergo segmental resection or total mastectomy on day 0.
Arm/Group | Treatment (MK2206) Dose Level 200mg | Treatment (MK2206) Dose Level 135mg | Treatment (MK2206) Dose Level 90mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (MK2206) Dose Level 200mg (N=4) | Treatment (MK2206) Dose Level 135mg (N=3) | Treatment (MK2206) Dose Level 90mg (N=5)
Fever (General disorders) | 1 | 0 | 0 — Participant also experienced Rash
Rash, Grade 3 (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (MK2206) Dose Level 200mg (N=4) | Treatment (MK2206) Dose Level 135mg (N=3) | Treatment (MK2206) Dose Level 90mg (N=5)
Mucositis, Grade 1 (Gastrointestinal disorders) | 1 | 0 | 1
Mucositis, Grade 2 (Gastrointestinal disorders) | 2 | 0 | 1
Rash, Grade 2 (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash, Grade 3 (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
Pruritus, Grade 1 (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus, Grade 3 (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Fever (General disorders) | 1 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less